CLINICAL TRIAL: NCT00740233
Title: Web-Based Survey of Pain, Stress and Complementary and Alternative Medicine
Acronym: PROCAIM
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Deborah Ackerman, University of California, Los Angeles
Other Study IDs: PROCAIM2008
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2009-02

CONDITIONS: Gastrointestinal Diseases; Chronic Pain; Stress; Anxiety; Depression
Keywords: fibromyalgia; irritable bowel syndrome; interstitial cystitis; chronic fatigue syndrome; vulvodynia; chronic stress; chronic pain; stress-related conditions; functional GI disorders
MeSH Terms: conditions — Gastrointestinal Diseases; Chronic Pain; Anxiety Disorders; Depression; Fibromyalgia; Irritable Bowel Syndrome; Cystitis, Interstitial; Fatigue Syndrome, Chronic; Vulvodynia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are inviting people with fibromyalgia, IBS, interstitial cystitis, chronic pain, and other chronic and recurring conditions to sign up and participate in a year-long Internet-based survey to study the effectiveness of alternative medicine and the interactions among stress and coping, pain, and treatment outcomes.

The survey is called PROCAIM, which stands for Patient-Reported Outcomes from Complementary, Alternative, and Integrative Medicine. PROCAIM was developed under a grant to UCLA researchers from the National Center for Complementary and Alternative Medicine.

This is a web-based study composed of surveys that will recur at intervals over 1 year!

TO ENROLL

* Log in to our web site: http://www.procaim.org/
* Register as a New User.
* Select clinic name: ClinicalTrials.gov.
* Read and sign the Consent Form.

After participants"sign" the form with their email address, participants can begin to answer the first in a series of questionnaires. The system will send participants email reminders at the time of each scheduled follow-up for one year.

For further information about PROCAIM, please contact:

* Deborah Ackerman, Ph.D.
* Department of Epidemiology
* UCLA School of Public Health
* Box 951772
* Los Angeles, CA 90095-1772
* deborah.ackerman@ucla.edu

DETAILED DESCRIPTION:
PROCAIM, which stands for Patient-Reported Outcomes from Complementary, Alternative, and Integrative Medicine, was developed to collect and manage longitudinal patient data and implement patient-based outcomes assessment protocols at clinical sites around the country that offer various forms of CAM as well as clinics that provide the combination of conventional medicine with complementary and alternative therapies. PROCAIM is currently being used for a 12 month longitudinal survey to evaluate interactions among stress, symptoms, severity, and general well-being among people with fibromyalgia, IBS, chronic fatigue, and other chronic pain conditions, and the frequency and impact of co-morbid conditions among users of complementary and alternative medicines.

ELIGIBILITY:
Inclusion Criteria:

* Everyone who has a computer and is fluent in English will be eligible.

Exclusion Criteria:

* Only people with access to personal computers and the Internet and fluency in English will be able to participate. These exclusions are not based on age, gender, pregnancy, racial, or ethnic origin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In general, participants will be: at least 18 years of age; ambulatory (i.e., not depending upon a wheelchair for mobility); and meet general criteria for psychosomatic or functional disorders including irritable bowel syndrome, other functional disorders, fibromyalgia, chronic pain, or related mood and anxiety disorders.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Perceived Stress, Mindfulness, Somatization | 1,3,6,9,12 months
  Online surveys at intervals over 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ackerman, Ph.D., Principal Investigator — UCLA School of Public Health